CLINICAL TRIAL: NCT00964743
Title: A Single Arm Pilot Study of Intrathecally Administered DepoCyt® With Systemic Sorafenib in the Treatment of Neoplastic Meningitis From Solid Tumors
Brief Title: Depocyt® With Sorafenib in Neoplastic Meningitis
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Low Accrual
Sponsor: H. Lee Moffitt Cancer Center and Research Institute (Other)
Collaborators: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MCC-15783; Bayer IST000266 (Other: Bayer)
Record Dates: First submitted 2009-08-24; First posted 2009-08-25 (Estimated); Results first posted 2012-04-19 (Estimated); Last update posted 2013-09-09 (Estimated); Status verified 2012-01

CONDITIONS: Neoplastic Meningitis
Keywords: Neurologic Oncology; Neoplastic Meningitis from solid tumors; Brain and Nervous System; Breast Cancer
MeSH Terms: conditions — Meningeal Carcinomatosis; Neurologic Manifestations; Breast Neoplasms | interventions — Sorafenib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Intrathecal DepoCyt and Oral Sorafenib (Experimental): This is a single arm pilot study. Investigators planned to enroll approximately 10 patients to receive concurrent intrathecal DepoCyt and oral Sorafenib. DepoCyt: through a reservoir every 2 weeks for 5 doses, then every 4 weeks for an additional 5 doses (a total of 10 DepoCyt treatments). Oral Sorafenib: at 400 mg twice a day throughout the treatment course until disease progression or death.
  Interventions: Drug: DepoCyt; Drug: Sorafenib

INTERVENTIONS:
Drug: DepoCyt — Patients were to receive DepoCyt through a reservoir every 2 weeks for 5 doses, then every 4 weeks for an additional 5 doses.
  Other Names: Liposomal Cytarabine; cytarabine liposome injection
Drug: Sorafenib — Patients received oral sorafenib at 400 mg twice a day
  Other Names: Nexavar; BAY 43-9006; oral multi-kinase inhibitor

SUMMARY:
The purpose of this study is to determine the tolerability and side effects of oral sorafenib in combination with intrathecal DepoCyt.

DETAILED DESCRIPTION:
After an Ommaya reservoir has been placed in the patient's head, the patient will receive DepoCyt through that reservoir every 2 weeks for 5 doses, then every 4 weeks for an additional 5 doses (a total of 10 DepoCyt treatments). Patients will also receive oral sorafenib at 400 mg twice a day throughout the treatment course until disease progression or death. Patients will receive brain magnetic resonance imaging (MRIs) with contrast (and whole spine, if necessary) and spinal fluid studies will be obtained every 8 weeks through the Ommaya reservoir until disease progression, death, or unacceptable toxicity. In addition, patients will have spinal fluid obtained to test for sorafenib levels at each study visit after the start of sorafenib as well as prior to sorafenib treatment for controls.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have neoplastic meningitis (NM) from solid tumor malignancy (excluding metastatic melanoma, leukemia, lymphoma, or primary malignant glioma) diagnosed by: Positive cerebrospinal fluid (CSF) cytology - or - Definitive neurologic signs/symptoms of NM with positive magnetic resonance imaging (MRI) findings or supportive CSF profile.
* Adequate bone marrow, liver, and renal function as assessed by the following: Hemoglobin ≥ 9.0 g/dl, Absolute neutrophil count (ANC) ≥ 1,500/mm³, Platelet count ≥ 100,000/mm³, Total bilirubin ≤ 1.5 times upper limit of normal (ULN), alanine transaminase (ALT) and aspartate transaminase (AST) ≤ 2.5 times the ULN ( ≤ 5 x ULN for patients with liver involvement), Creatinine ≤ 1.5 times ULN, international normalized ratio (INR) < 1.5 or a prothrombin time/partial thromboplastin time (PT/PTT) within normal limits. Patients receiving anti-coagulation treatment with an agent such as warfarin or heparin may be allowed to participate. For patients on warfarin, the international normalized ratio (INR) should be measured prior to initiation of sorafenib and monitored at least weekly, or as defined by the local standard of care, until INR is stable
* Must have a Karnofsky performance score ≥ 60% (i.e. the patient must be able to care for himself/herself with occasional help from others)
* Must be healthy enough to receive ventricular access device (VAD) placement.
* Patients with a ventriculoperitoneal (VP) shunt that have an on/off device in their shunt systems are eligible for the study provided they are able to tolerate shunt closure for ≥ 4 hours without developing clinical signs of increased intracranial pressure.
* Women of childbearing potential (WOCBP) must have a negative serum pregnancy test performed within 7 days prior to the start of treatment
* WOCBP and men must agree to use adequate contraception (barrier method of birth control) prior to study entry and for the duration of study participation. Men should use adequate birth control for at least 3 months after the last administration of sorafenib.
* Ability to understand and the willingness to sign a written informed consent. A signed informed consent must be obtained prior to any study specific procedures.

Exclusion Criteria:

* Neoplastic meningitis (NM) from metastatic melanoma, leukemia, lymphoma, or primary malignant glioma
* Uncontrolled systemic disease from their primary cancer
* Must not have had prior intrathecal chemotherapy, sorafenib, or brain or spine radiation for the treatment of neoplastic meningitis.
* Concomitant therapy with high-dose systemic methotrexate, cytarabine, thiotepa, or an agent known to have penetration into the central nervous system (CNS)
* Patients with clinical evidence of obstructive hydrocephalus or compartmentalization of CSF flow as documented by radioisotope Indium (Technetium-DTPA when Indium unavailable) flow study are not eligible for this trial. If patients have evidence of cerebrospinal fluid (CSF) flow blockage that is subsequently proven to be relieved after focal radiation therapy (XRT), they can enroll immediately after repeat flow study shows block to be relieved.
* Use of any investigational drug within 28 days prior to study entry.
* Patients with a life expectancy of ≤ 2 months
* Cardiac disease: Congestive heart failure > class II New York Heart Association (NYHA). Must not have unstable angina or new onset angina (began within the last 3 months)or myocardial infarction within past 6 months.
* Cardiac ventricular arrhythmias requiring anti-arrhythmic therapy.
* Uncontrolled hypertension defined as systolic blood pressure > 150 mmHg or diastolic pressure > 90 mmHg, despite optimal medical management.
* Known human immunodeficiency virus (HIV) infection or chronic Hepatitis B or C.
* Active clinically serious infection > Common Terminology Criteria for Adverse Events (CTCAE) Grade 2.
* Thrombolic or embolic events such as a cerebrovascular accident including transient ischemic attacks within past 6 months.
* Pulmonary hemorrhage/bleeding event ≥ CTCAE Grade 2 within 4 weeks of first dose of study drug.
* Any other hemorrhage/bleeding event ≥ CTCAE Grade 3 within 4 weeks of first dose of study drug.
* Serious non-healing wound, ulcer, or bone fracture.
* Evidence or history of bleeding diathesis or coagulopathy
* Major surgery, open biopsy or significant traumatic injury within 4 weeks of first study drug.
* Use of St. John's Wort or rifampin.
* Known or suspected allergy to sorafenib or any agent given in the course of this trial.
* Any condition that impairs patient's ability to swallow whole pills.
* Any malabsorption problem.
* Patients who are pregnant or breast-feeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2009-08; Primary Completion 2011-02 (Actual); Study Completion 2011-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Edward Pan, M.D., Principal Investigator — H. Lee Moffitt Cancer Center and Research Institute
Locations (1):
- H. Lee Moffitt Cancer Center and Research Institute, Tampa, Florida, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Intrathecal DepoCyt and Oral Sorafenib
Started | 2
Completed | 0
Not Completed | 2
Not completed — Neither patient completed 8 weeks of tre | 2

BASELINE CHARACTERISTICS:
Arm/Group | Intrathecal DepoCyt and Oral Sorafenib
Number analyzed (Participants) | 2
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 0
  >=65 years | 2
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 1
Region of Enrollment [Number; unit: participants]
  United States | 2

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Events (AEs)
Description: Safety and tolerability of sorafenib with DepoCyt. Toxicities were to be reported using tables and descriptive statistics by type and grade. All patients were to be followed up until death.
Time Frame: 6 Months
Population: All participants
Measure: Number; unit: participants
Arm/Group | Intrathecal DepoCyt and Oral Sorafenib
Number analyzed (Participants) | 2
participants | 2

2. Secondary Outcome: Number of Participants With Progression Free Survival (PFS) at 6 Months
Description: Kaplan-Meier analysis of PFS was to be performed and the PFS at 6 months in the study patients were be empirically described. All patients were to be followed up until death.
Time Frame: 6 Months
Population: The study closed early due to low accrual of 2 of 10 expected patients. Neither patient completed 8 weeks of treatment as outlined in the protocol. Both patients expired before reaching the 6 month Progression Free Survival endpoint.
Arm/Group | Intrathecal DepoCyt and Oral Sorafenib
Number analyzed (Participants) | 0

3. Secondary Outcome: Number of Participants With Overall Survival (OS)
Description: Several secondary endpoints were to be analyzed in a descriptive fashion. All patients were to be followed up until death.
Time Frame: 6 Months
Population: as for outcome 2
Arm/Group | Intrathecal DepoCyt and Oral Sorafenib
Number analyzed (Participants) | 0

4. Secondary Outcome: Sorafenib Levels in Cerebrospinal Fluid (CSF)
Description: CSF sorafenib level was to be measured over time, and the means and standard errors of the sorafenib level were to be plotted at specific sampling time points. CSF sorafenib levels may also have been correlated with patients' PFS, OS, or cytology using descriptive statistical methods (e.g., KM analysis stratified by high vs. low CSF sorafenib levels). The log transformation of lab values were to be employed on the continuous variables whenever necessary.
Time Frame: 6 Months
Population: as for outcome 2
Arm/Group | Intrathecal DepoCyt and Oral Sorafenib
Number analyzed (Participants) | 0

5. Secondary Outcome: CSF and Serum Vascular Endothelial Growth Factor (VEGF) Levels
Description: CSF and serum VEGF levels were to be measured over time, and the means and standard errors of the respective VEGF levels were to be plotted at specific sampling time points. The respective VEGF levels may also have been correlated with patients' PFS, OS, or cytology using descriptive statistical methods similarly as mentioned above. The log transformation of lab values were to be employed on the continuous variables whenever necessary.
Time Frame: 6 Months
Population: as for outcome 2
Arm/Group | Intrathecal DepoCyt and Oral Sorafenib
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: 8 months
Description: First On Study (9/10/09) to last Off Study (5/18/10)
Arm/Group | Intrathecal DepoCyt and Oral Sorafenib
Serious Adverse Events (participants affected / at risk) | 2/2
Other Adverse Events (participants affected / at risk) | 1/2
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Intrathecal DepoCyt and Oral Sorafenib (N=2)
Death not associated with CTCAE term - Death not otherwise specified (NOS) (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) — Death occurred within 30 days. Unrelated to study treatment. Death not associated with Common Terminology Criteria for Adverse Events (CTCAE)
Death not associated with CTCAE term - Disease progression not otherwise specified (NOS) (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) — Death occurred within 30 days. Unrelated to study treatment. Death not associated with Common Terminology Criteria for Adverse Events (CTCAE)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Intrathecal DepoCyt and Oral Sorafenib (N=2)
Hemoglobin (Blood and lymphatic system disorders) | 1 (1) — Grade 1. Unrelated.
Hypotension (Cardiac disorders) | 1 (1) — Grade 1. Unrelated.
Fever (in the absence of neutropenia, where neutropenia is defined as ANC <1.0 x 10^9/L (General disorders) | 1 (1) — Grade 1. Unrelated. Fever (in the absence of neutropenia, where neutropenia is defined as absolute neutrophil count (ANC) <1.0 x 10^9/L
Ulceration (Skin and subcutaneous tissue disorders) | 1 (1) — Grade 2. Unrelated.
Anorexia (Gastrointestinal disorders) | 1 (1) — Grade 2. Unrelated.
Dehydration (Gastrointestinal disorders) | 1 (1) — Grade 2. Unrelated.
Infection with unknown ANC-Mucosa (Infections and infestations) | 1 (1) — Grade 1. Unrelated. Infection with unknown absolute neutrophil count (ANC)-Mucosa
Edema: limb (Blood and lymphatic system disorders) | 1 (1) — Grade 2. Unrelated.
Somnolence/depressed level of consciousness (Nervous system disorders) | 1 (1) — Grade 1. Unrelated
Cognitive disturbance (Nervous system disorders) | 1 (1) — Grade 3. Unrelated.

LIMITATIONS AND CAVEATS:
The study closed early due to low accrual of 2 of 10 expected patients. Neither patient completed 8 weeks of treatment as outlined in the protocol. Both patients expired before reaching the 6 month Progression Free Survival endpoint.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes